CLINICAL TRIAL: NCT07120880
Title: Efficacy of a Combination of Chronotherapeutics for the Treatment of Major Depressive Episode (MDE) With Insomnia: a Multicenter, Randomized, 2*2 Factorial, Double-blind, Placebo-controlled Trial
Brief Title: Efficacy of Chronotherapeutic Combination for Major Depressive Episode With Insomnia
Acronym: CombiChronoS
Status: Not yet recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: Double | Purpose: Treatment
Other Study IDs: APHP230869
Record Dates: First submitted 2025-07-11; First posted 2025-08-13 (Actual); Last update posted 2025-08-13 (Actual); Status verified 2025-07

CONDITIONS: Major Depressive Disorder (MDD) With Insomnia
Keywords: Major depressive episode; Insomnia; Light therapy; Melatonin
MeSH Terms: conditions — Depressive Disorder, Major; Sleep Initiation and Maintenance Disorders | interventions — SHORT ROOT protein, Arabidopsis

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- A (Active Comparator): Patients receiving active light therapy (approx. 10,000 Lux) and prolonged-release melatonin 2 mg taken 1 hour before bedtime, in combination with sleep and hygiene rules (SHR) and antidepressant treatment (AD)
  Interventions: Procedure: AD + SHR + active LT and extended-release melatonin 2mg
- B (Active Comparator): Patients receiving active light therapy (approx. 10,000 Lux) and placebo melatonin, in combination with SHR and AD.
  Interventions: Procedure: AD + SHR + active LT and placebo melatonin
- C (Active Comparator): Patients receiving placebo light therapy (filtered to approx. <10 Lux) and prolonged-release melatonin 2 mg taken 1 hour before bedtime, in combination with SHR and AD.
  Interventions: Procedure: AD + SHR + placebo LT and extended-release melatonin 2mg
- D (Placebo Comparator): Patients receiving placebo light therapy (filtered to approx. <10 Lux) and placebo melatonin (control group), in combination with SHR and AD.
  Interventions: Procedure: AD + SHR + placebo LT and placebo melatonin

INTERVENTIONS:
Procedure: AD + SHR + active LT and extended-release melatonin 2mg — Patients will receive an SSRI antidepressant (e.g., Fluoxetine, Sertraline, Paroxetine, Escitalopram) or SNRI (e.g., Venlafaxine, Duloxetine) antidepressant (as clinically appropriate), combined with sleep hygiene education, daily morning LT (10,000 lux for 30 minutes between 7-8 a.m. using the Dayvia Slim Style 3 lamp), and 2 mg of extended-release melatonin taken one hour before bedtime, all for a duration of 8 weeks.
  Arms: A
Procedure: AD + SHR + active LT and placebo melatonin — Patients will receive an SSRI or SNRI, sleep hygiene instructions, daily morning bright LT (10,000 lux, 30 cm, 30 min, 7-8 a.m., using Dayvia Slim Style 3 lamps), and placebo melatonin taken one hour before bedtime, all for a duration of 8 weeks.
  Arms: B
Procedure: AD + SHR + placebo LT and extended-release melatonin 2mg — Patients will receive an SSRI or SNRI, sleep hygiene instructions, daily placebo light exposure (<10 lux, 30 cm, 30 min, 7-8 a.m., using Dayvia Slim Style 3 lamps in non-therapeutic mode), and 2 mg of extended-release melatonin taken one hour before bedtime, all for a duration of 8 weeks.
  Arms: C
Procedure: AD + SHR + placebo LT and placebo melatonin — Patients will receive an SSRI or SNRI, sleep hygiene instructions, daily placebo light exposure (<10 lux, 30 cm, 30 min, 7-8 a.m., using Dayvia Slim Style 3 lamps), and oral placebo melatonin taken one hour before bedtime, all for a duration of 8 weeks.
  Arms: D

SUMMARY:
Major Depressive Disorder (MDD) affects 5% of the global population and is the second leading cause of disability worldwide. Despite the widespread use of antidepressants, 50-60% of patients do not respond adequately after 8 weeks of treatment. Insomnia, present in approximately 85% of individuals with MDD, is a frequent and persistent symptom that contributes to poor treatment outcomes. Targeting insomnia has been shown to enhance both symptom remission and functional recovery. In this context, combined therapeutic strategies are often used to optimize the antidepressant response. Among them, chronotherapeutic approaches, such as light therapy and prolonged-release melatonin, have demonstrated rapid antidepressant effects and are beneficial in regulating sleep and circadian rhythms. Light therapy shows an efficacy comparable to antidepressants and, when used in combination with them, can double treatment effectiveness. Melatonin is also recommended in the management of depression-related insomnia. This multicenter, randomized, double-blind, placebo-controlled trial with a 2x2 factorial design aims to evaluate the efficacy of two chronotherapeutic interventions, 8 weeks of active light therapy and 2 mg of prolonged-release melatonin-administered alone or in combination, on depressive symptom reduction at 8 weeks in adult patients with MDD and comorbid insomnia. The primary outcome is the change in Montgomery-Åsberg Depression Rating Scale (MADRS) score from baseline to week 8. All participants will receive antidepressant treatment and sleep hygiene education. This study proposes a novel therapeutic strategy combining pharmacological and non-pharmacological interventions to address both depression and insomnia, with the goal of improving outcomes, especially for the 40% of patients who do not adequately respond to antidepressants alone.

DETAILED DESCRIPTION:
Major Depressive Disorder (MDD) affects approximately 5% of the global population and represents the second leading cause of disability worldwide. Despite the availability of pharmacological treatments, particularly antidepressants, their efficacy remains limited: nearly 50 to 60% of patients do not respond adequately after 8 weeks of treatment. One of the most common and persistent symptoms in MDD is insomnia, which affects about 85% of patients and frequently persists even after partial improvement of mood symptoms. Insomnia is not only a residual symptom but also a marker of poor prognosis and treatment resistance. Addressing sleep disturbances directly has been shown to enhance both symptomatic and functional remission in depression, making it a promising target for intervention.

In clinical practice, combination strategies are increasingly employed to improve therapeutic response, particularly in patients who are only partially responsive to antidepressant medication. Among these strategies, chronotherapeutic interventions, such as light therapy and prolonged-release melatonin, offer a compelling approach. These treatments have demonstrated rapid antidepressant effects, with some studies reporting clinical improvements as early as the first week of treatment. Additionally, both interventions are known to positively influence sleep quality and circadian rhythm regulation, which are often disrupted in depressive disorders.

Light therapy (LT), in particular, has shown efficacy comparable to that of antidepressants and works by synchronizing the sleep-wake cycle. When used in combination with antidepressants, LT has been associated with significantly greater reductions in depressive symptoms than antidepressants alone. Similarly, prolonged-release melatonin has been recommended in the management of insomnia comorbid with depression, further supporting the rationale for combining these chronotherapeutic agents.

This study is a multicenter, randomized, double-blind, placebo-controlled trial designed in a 2x2 factorial format. It aims to evaluate the efficacy of two chronotherapeutic interventions, active light therapy (10,000 lux) for 8 weeks and 2 mg prolonged-release melatonin for 8 weeks, administered alone or in combination, in improving depressive symptoms at 8 weeks. The trial will enroll adult patients diagnosed with moderate to severe MDD and comorbid insomnia. The primary objective is to assess the change in depressive symptom severity, measured by the Montgomery-Åsberg Depression Rating Scale (MADRS) score, from baseline to week 8.

All participants, regardless of group allocation, will receive standard antidepressant treatment and structured sleep hygiene counseling to ensure a consistent baseline of care. This approach reflects real-world practices and enhances the ecological validity of the trial. The study also incorporates objective and subjective measures of sleep and circadian rhythms to explore the broader impact of the interventions.

By evaluating the combined and individual effects of light therapy and melatonin alongside standard care, this study seeks to establish an innovative and comprehensive therapeutic model. The goal is to improve outcomes for individuals with MDD and insomnia, particularly the substantial proportion of patients, up to 40%, who do not achieve adequate response with antidepressants alone. This trial represents a significant step toward more personalized, effective, and integrated treatment strategies for depression.

ELIGIBILITY:
Inclusion Criteria:

1. Adults aged between 18 and 65 years (to avoid the risk of cataract associated with light therapy) with a diagnosis of a major depressive episode (MDE) in the context of unipolar depression (according to DSM-5 criteria).
2. Diagnosis of comorbid insomnia with the MDE, defined by difficulty initiating sleep, and/or maintaining sleep, and/or early morning awakenings with daytime consequences, occurring at least three times per week (according to DSM-5 and ICSD-3, in line with European guideline recommendations).
3. Outpatients or inpatients treated for MDE in one of the psychiatric departments of the study centers, or in the sleep medicine department, for a minimum treatment duration of 8 weeks.
4. Patients not currently receiving antidepressant treatment for the current MDE (previous use of antidepressants is allowed, provided treatment was stopped at least one month prior to study participation).
5. A MADRS score ≥ 20 (clinician-rated), indicating at least a moderate-intensity depressive episode.
6. An ISI score ≥ 8 (clinician-rated), indicating at least mild and clinically significant insomnia.
7. No exposure to light therapy in the month prior to inclusion.
8. Ability to understand and sign the informed consent form.
9. Use of highly effective contraception for women of childbearing potential.

Exclusion Criteria:

1. Individuals under legal guardianship or deprived of liberty
2. Ophthalmologic conditions (e.g., cataract, glaucoma, age-related macular degeneration) or diseases affecting the retina (e.g., retinitis pigmentosa, diabetes, herpes, etc.)
3. The following disorders (according to DSM-5): schizophrenia and other psychotic disorders; bipolar disorder, particularly (hypo)manic episodes (YMRS score ≥ 12); other unstable mental disorders
4. Other unstable general medical conditions
5. Pregnant or breastfeeding women
6. Hypersomnia with prolonged total sleep time secondary to the depressive episode, according to ICSD-3 criteria
7. Current depressive episode already being treated with an antidepressant
8. Presence of a high suicidal risk, as assessed by the Columbia-Suicide Severity Rating Scale (C-SSRS, score ≥ 4)
9. Ongoing melatonin treatment at the time of inclusion

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 184 (Estimated)
Dates: Start 2025-09 (Estimated); Primary Completion 2028-05 (Estimated); Study Completion 2029-05 (Estimated)

PRIMARY OUTCOMES:
Assessment of the efficacy of two chronotherapeutics (LT and extended-release melatonin 2mg), alone or combined, associated to AD on depressive symptoms reduction after 8 weeks of treatment | At baseline (Week 0) and at Week 8
  Measure the change in Montgomery-Åsberg Depression Rating Scale (MADRS) total score between the inclusion visit (V0, S0) and Week 8 (V3, S8) in patients with moderate to severe major depressive episode and insomnia

SECONDARY OUTCOMES:
Assessment of the efficacy of chronotherapeutics, combine or alone, on depressive symptoms evolution | Weeks 1, 4, 8, and Month 3
  Measure changes in MADRS scores from baseline (inclusion visit) to each follow-up visit (Week 1, Week 4, Week 8, and Month 3).
Determination of the rate of therapeutic response to chronotherapeutics at each follow-up visit | Weeks 1, 4, 8, and Month 3
  Proportion of patients achieving ≥50% reduction in MADRS score at each follow-up visit (Week 1, Week 4, Week 8 and Month 3) as compared to baseline (inclusion visit)
Determination of the rate of remission in depressive symptoms | Weeks 4, 8, and Month 3
  Proportion of patients with MADRS score ≤10 at specified time points (Weeks 4, 8 and Month 3).
Evaluation of the impact of chronotherapeutics on subjective sleep | Weeks 1, 4, 8, and Month 3
  Assessment using self-reported sleep questionnaires, sleep-wake rhythm diaries, and sleep logs
Evaluation of the impact of chronotherapeutics on circadian rhythm | Weeks 1, 4, 8, and Month 3
  Assessment using self-reported sleep questionnaires, sleep-wake rhythm diaries, and sleep logs
Evaluation of changes in objective sleep measured by actigraphy | Weeks 1, 4, and 8
  Total sleep time
Evaluation of changes in objective sleep measured by actigraphy | Weeks 1, 4, and 8
  Wake After Sleep Onset (WASO)
Evaluation of changes in objective sleep measured by actigraphy | Weeks 1, 4, and 8
  Fragmentation index
Evaluation of changes in objective sleep measured by actigraphy | Weeks 1, 4, and 8
  Sleep efficiency
Evaluation of changes in objective sleep measured by actigraphy | Weeks 1, 4, and 8
  Time in bed
Evaluation of changes in sleep rhythm parameters measured by actigraphy | Weeks 1, 4, and 8
  Total Sleep Time
Evaluation of changes in sleep rhythm parameters measured by actigraphy | Weeks 1, 4, and 8
  Wake After Sleep Onset (WASO)
Evaluation of changes in sleep rhythm parameters measured by actigraphy | Weeks 1, 4, and 8
  Fragmentation Index
Evaluation of changes in sleep rhythm parameters measured by actigraphy | Weeks 1, 4, and 8
  Sleep Efficiency
Evaluation of changes in sleep rhythm parameters measured by actigraphy | Weeks 1, 4, and 8
  Time in Bed
Evaluation of changes in objective actigraphy-derived sleep and rhythm parameters | Weeks 1, 4, and 8
  Relative amplitude
Evaluation of changes in objective actigraphy-derived sleep and rhythm parameters | Weeks 1, 4, and 8
  Interdaily stability/variability
Evaluation of changes in objective actigraphy-derived sleep and rhythm parameters | Weeks 1, 4, and 8
  L5/M10 onset markers
Modeling of the longitudinal trajectory of MADRS scores | From baseline to Week 8 and from baseline to Month 3
  Analyze the slope of MADRS score changes across visits to characterize symptom progression or improvement.
Measurement of time to therapeutic response | From baseline to Month 3
  Time (in days) from inclusion to achievement of ≥50% reduction in MADRS score.
Evaluation of the tolerability of chronotherapeutic combinations | Weeks 1, 4, and 8
  Evaluate adverse events using the PRISE-M side effects questionnaire.
Evaluation of mood state | Weeks 1, 4, 8, and Month 3
  Scores on YMRS (mania)
Evaluation of mood state | Weeks 1, 4, 8, and Month 3
  C-SSRS (suicidal ideation)
Evaluation of mood state | Weeks 1, 4, 8, and Month 3
  QIDS-SR (depression)
Evaluation of mood state | Weeks 1, 4, 8, and Month 3
  GAD-7 (anxiety)
Evaluation of mood state | Weeks 1, 4, 8, and Month 3
  CGI (clinical global impression)
Evaluation of global functioning evolution | Weeks 1, 4, 8, and Month 3
  Scores on YMRS (mania)
Evaluation of global functioning evolution | Weeks 1, 4, 8, and Month 3
  C-SSRS (suicidal ideation)
Evaluation of global functioning evolution | Weeks 1, 4, 8, and Month 3
  QIDS-SR (depression)
Evaluation of global functioning evolution | Weeks 1, 4, 8, and Month 3
  GAD-7 (anxiety)
Evaluation of global functioning evolution | Weeks 1, 4, 8, and Month 3
  CGI (clinical global impression)

CONTACTS AND LOCATIONS:
Overall Officials: Pierre-Alexis GEOFFROY, Pr, Principal Investigator — Assistance Publique Hopitaux de Paris
Locations (1):
- Hôpital Bichat-Claude Bernard, Paris, France

IPD SHARING:
Plan to Share IPD: No